CLINICAL TRIAL: NCT06834503
Title: Bioequivalence Study of Clonazepam 2 Mg Tablets/immediate Release Tablets in Healthy Subjects in a Fasting Condition
Brief Title: Bioequivalence Study of Clonazepam 2 Mg Tablets
Acronym: Clonazepam
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Atencion e Investigacion Medica (Network)
Responsible Party: Principal Investigator, Humberto Reynales MD MSc PhD, Principal Investigator, Centro de Atencion e Investigacion Medica
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CLONAZ-BIO-002-2023
Record Dates: First submitted 2025-01-29; First posted 2025-02-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Healthy Donors
MeSH Terms: interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Period 1 (Active Comparator): Rivotril® 2 mg
  Interventions: Drug: Rivotril®
- Period 2 (Active Comparator): Clonazepam TQ 2 mg
  Interventions: Drug: Clonazepam TQ 2 mg

INTERVENTIONS:
Drug: Rivotril® — Rivotril® 2 mg
  Arms: Period 1
Drug: Clonazepam TQ 2 mg — Test
  Arms: Period 2

SUMMARY:
Demonstrate the bioequivalence in 1 study, in fasting condition of two formulations of clonazepam 2 mg Tablets / tablets immediate release in order to establish that there are no significant pharmacokinetic differences.

DETAILED DESCRIPTION:
To establish the main pharmacokinetic variables of the two formulations.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 18 and 50 years of age at the time of signing the informed consent form.
* Women who are not capable of conceiving (To be considered not capable of conceiving she must be at least 1 year postmenopausal or surgically sterile) or who are not pregnant or breastfeeding.
* Women of childbearing capacity must be using adequate contraception for the past 6 months and agree to continue using adequate contraception for 30 days after signing the consent form.
* Have been clinically diagnosed as healthy by the study physician.
* Subjects with the clinical laboratory results requested in the protocol (Table 2) within normal ranges and/or fit by medical selection. Current for 3 months.
* Subjects non-smokers for the last 3 months at the time of signing the informed consent.
* Having signed the informed consent for the study.
* Subjects sexually active or of reproductive age must use an effective contraceptive method during and for at least 7 days after the end of the study.
* Body mass index between 18-30 kg/m2 at the time of inclusion in the study.
* Subject with complete contact information (cell phone and/or landline contact, address).
* Subject with a family member or guardian with a contact telephone number.
* Subject with the availability of time to comply with the scheduled visits and activities.
* Subject willing to comply with the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Subject with a diagnosis of renal, cardiac, hepatic, immunological, dermatological, endocrine, gastrointestinal, neurological or psychiatric disease, compulsive depressive disorder.
* Subject with diagnosis of hematological disorders, such as anemias and/or polycythemia.
* Subjects with history of gastric surgeries.
* Permanent or temporary use during the last 5 days prior to the administration of the investigational product of the study of any type of medication either on their own initiative or by medical prescription. Except female patients who are planning regularly with the same contraceptive method in the last 6 months prior to the start of the present study.
* Pregnant or breastfeeding women (Table 2).
* Xanthine consumption from coffee, tea or chocolate during the 48 hours prior to hospitalization.
* Alcohol consumption of more than 16 g per week equivalent to 1 beer or 2 glasses of wine during the 5 days prior to administration of the investigational product.
* Positive test for consumption of drugs of abuse or psychoactive substances at the time of screening or prior to administration of the investigational product. (Table 2)
* Known hypersensitivity to the active substance or excipients of the test product.
* Medical history of angioedema or anaphylaxis.
* Subject diagnosed with human immunodeficiency virus, hepatitis B (surface antigen) or hepatitis C (surface antigen) positive infection.
* Having participated in clinical trials in the 4 months prior to the time of signing the informed consent.
* Have donated blood or reported blood loss greater than 500 mL in the 30 days prior to the time of investigational product administration.
* Subject with clinically significant acute illness or temperature > 38°C within 24 hours prior to administration of the investigational product.
* Subject with any contraindication to blood collection due to bleeding disorders or thrombocytopenia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures | 0 - 72 Hours
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic Outcome Measures | 0 - 6 Hours
  The plasma concentration max

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Measures | 0 - 6 Hours
  tmax .

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Nov 2025 Dic 2030
Access Criteria: Indicate whether a proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed
URL: https://www.caimed.com/